CLINICAL TRIAL: NCT03280030
Title: A Phase II, Randomized, Double-blind, Multi-center, Placebo-controlled Study to Evaluate the Efficacy and Safety of Twice Daily Oral Midostaurin in Combination With Daunorubicin/Cytarabine Induction, High-dose Cytarabine Consolidation, and Midostaurin Single Agent Continuation Therapy in Newly Diagnosed Patients With FLT3-mutated Acute Myeloid Leukemia (AML).
Brief Title: A Study of Midostaurin Efficacy and Safety in Newly Diagnosed Patients With FLT3-mutated AML
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CPKC412A2220
Record Dates: First submitted 2017-09-08; First posted 2017-09-12 (Actual); Results first posted 2025-02-11 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Acute Myeloid Leukemia
Keywords: midostaurin; PKC412; cytarabine; daunorubicin; acute myeloid leukemia; combination treatment; FLT3; acute myeloid leukemia (AML); acute myelogenous leukemia (AML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — midostaurin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Midostaurin (Experimental): Patients took study drug on day 8-21 during induction and consolidation phase; then on days 1-28 for 12 cycles in the continuation (post consolidation) phase.
  Interventions: Drug: Midostaurin
- Placebo (Placebo Comparator): Patients took placebo on day 8-21 during induction and consolidation phase; then on days 1-28 for 12 cycles in the continuation (post consolidation) phase.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Midostaurin — Midostaurin 50 mg [two 25 mg capsules] were administered twice per day by mouth on day 8-21 during induction and consolidation phase; then on days 1-28 for 12 cycles in the continuation (post consolidation) phase.
  Other Names: PKC412
  Arms: Midostaurin
Drug: Placebo — Placebo, two capsules, were administered twice per day by mouth on day 8-21 during induction and consolidation phase; then on days 1-28 for 12 cycles in the continuation (post consolidation) phase.
  Arms: Placebo

SUMMARY:
This study evaluated the efficacy and safety of midostaurin in combination with daunorubicin/cytarabine induction, high dose cytarabine consolidation and midostaurin single agent continuation therapy in newly diagnosed patients with FLT3-mutated acute myeloid leukemia (AML).

DETAILED DESCRIPTION:
This was a Phase II, multi-center trial consisting of two parts; Part 1: an open label, safety evaluation part in Japan only (minimum of three evaluable subjects) and Part 2: a double-blind, randomized, placebo-controlled part (60 subjects). Part 1 in Japan and Part 2 outside Japan were initiated simultaneously. Part 1 was conducted to evaluate the safety and tolerability of midostaurin in combination with daunorubicin/cytarabine induction and high-dose cytarabine consolidation in Japanese subjects and was a pre-requisite before allowing participation of Japan in Part 2. Data from Part 1 was reviewed by an Independent safety Committee (ISC) designated by the Sponsor. The ISC reviewed all available safety data in subjects from Japan up to the time of the safety review data cut-off date (6-Sep-2018). A meeting with the ISC was held on 25-Sep-2018: based on safety evaluation in three evaluable subjects, the ISC members recommended to start Part 2 in Japan.

Part 2 of the study included screening phase, treatment phase composed of up to 18 cycles of midostaurin/placebo treatment in combination with chemotherapy (daunorubicin and cytarabine) during induction and consolidation and alone during continuation and 30 days safety follow up from last dose of study treatment (daunorubicin or cytarabine or midostaurin/placebo); and follow up phase for continued remission and survival follow-up (until 36 months after Day 1 of the last subject). Subjects who provided written informed consent were screened for eligibility during the period up to 7 days immediately prior to starting chemotherapy (Day 1). The subject was randomized at Day 8 to receive either midostaurin or placebo only if FLT3 status was mutated. Treatment phase included induction, consolidation and continuation therapies.

Induction therapy: All screened subjects started induction therapy with chemotherapy from Day 1 to Day 7, while the FLT3 mutation status was being determined. Subjects who achieved CR already with induction Cycle 1 went directly to consolidation therapy without a second cycle of induction therapy. Subjects who did not achieve CR with one cycle of induction received a second induction cycle with same treatment as in Cycle 1. Subjects who did not achieve CR after induction 2 discontinued the study treatment and were followed in safety follow up and survival follow-up.

Consolidation therapy: Subjects who achieved a CR after 1 or 2 cycles of induction received consolidation therapy with 3 cycles of high-dose cytarabine for the Japan Adult Leukemia Study Group (JALSG) regimen and 4 cycles of high-dose cytarabine as tolerated for the Randomized AML Trial In FLT3+ subjects <60 Years old (RATIFY) regimen. Subjects received midostaurin/placebo, orally twice a day, on Days 8 to 21 of each cycle. Each consolidation cycle began within two weeks following hematopoietic recovery (ANC ≥ 1.0 x 109/L, platelet count ≥ 100 x 109/L) but no sooner than four weeks from the beginning of the previous cycle.

Continuation therapy: After hematopoietic recovery (ANC ≥ 1.0 x 109/L, platelet count ≥ 100 x 109/L) following the final cycle of consolidation but no sooner than 14 days after the last dose of midostaurin/placebo during the last consolidation cycle, subjects who maintained a CR received up to 12 cycles (28 days/cycle) of continuous therapy with midostaurin or placebo twice a day. Safety was assessed in this treatment phase for each subject until 30 days after the end of treatment (EOT) and included routine safety monitoring.

The follow-up phases included post treatment follow-up and survival follow-up. During post-treatment follow-up, all subjects continued to be assessed for relapse i.e. every 2 months during years 1 and 2, every 3 months on year 3 and 4 and then yearly and at time of relapse until relapse, withdrawal of consent, death, loss to follow up, or end of study, whichever was earlier following the end of study treatment for any reason other than persistent AML. Subjects who discontinued study treatment due to persistent AML or relapse and the post treatment follow-up phase due to relapse entered a survival follow-up period during which survival was recorded every 3 months. Survival information was obtained by clinical visits or telephone calls or other means until death, withdrawal of consent, lost to follow-up or end of study, whichever was earlier.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AML (≥ 20% blasts in the bone marrow based on WHO 2016 classification). Patients with APL (acute promyelocytic leukemia) with PML-RARA are not eligible
* Documented presence of an ITD and/or TKD activating mutation in the FLT3 gene, as determined by analysis in a Novartis designated laboratory An exception will be patients who are enrolled into the part 1 in Japan, who may be treated with midostaurin irrespective of AML FLT3 genotype.
* Patients must meet the following laboratory value criteria that indicate adequate organ function at the screening visit:

  * Estimated creatinine clearance ≥ 30 ml/min
  * Total bilirubin ≤ 1.5 x ULN, except in the setting of isolated Gilbert syndrome
  * Aspartate transaminase (AST) ≤ 3.0 x ULN
  * Alanine transaminase (ALT) ≤ 3.0 x ULN
* Suitability for intensive chemotherapy in the judgment of the investigator

Exclusion Criteria:

* Neurologic symptoms suggestive of CNS leukemia unless CNS leukemia has been excluded by a lumbar puncture. Patients with CSF fluid positive for AML blasts are not eligible
* Developed therapy-related AML after prior radiotherapy (RT) or chemotherapy for another cancer or disorder
* Known hypersensitivity to midostaurin, cytarabine or daunorubicin or to any of the excipients of midostaurin/placebo, cytarabine or daunorubicin
* Abnormal chest X-ray unless the abnormality represents a non-active, or non-clinically significant finding, such as scarring (subjects with controlled non active lung infection are eligible)
* Known impairment of gastrointestinal (GI) function or GI disease that might alter significantly the absorption of midostaurin
* Cardiac or cardiac repolarization abnormality
* Pregnant or nursing (lactating) women
* Women of child-bearing potential, unless they are using highly effective methods of contraception during dosing and for 4 months after stopping medication

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2018-04-06 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2022-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (32):
- Novartis Investigative Site, Pokfulam, Hong Kong
- Japan (22):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Toyoake, Aichi-ken
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Fukushima, Fukushima
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Isehara, Kanagawa
  - Novartis Investigative Site, Nagasaki, Nagasaki
  - Novartis Investigative Site, Okayama, Okayama-ken
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Ōsaka-sayama, Osaka
  - Novartis Investigative Site, Hamamatsu, Shizuoka
  - Novartis Investigative Site, Shimotsuke, Tochigi
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Shinagawa Ku, Tokyo
  - Novartis Investigative Site, Aomori
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Kochi
  - Novartis Investigative Site, Kyoto
  - Novartis Investigative Site, Osaka
  - Novartis Investigative Site, Yamagata
- Russia (2):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
- South Korea (2):
  - Novartis Investigative Site, Seoul, Seocho Gu
  - Novartis Investigative Site, Seoul
- Taiwan (4):
  - Novartis Investigative Site, Putzu City, Chiayi Hsien
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
- Novartis Investigative Site, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1837

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Part 1 of the study enrolled 5 Japan adult subjects with newly diagnosed (ND) FLT3-mutated or non-mutated AML. Part 2 randomized 62 adult subjects with ND FLT3-mutated AML. The efficacy analysis was on the 62 randomized subjects in Part 2. The safety analysis was considered separately on 5 subjects in Part 1 & 61 out of 62 randomized subjects in Part 2, as 1 subject did not receive randomized treatment (placebo). The PK analysis was on subjects treated with midostaurin in Part 1 or Part 2.
Pre-assignment Details: Subjects were enrolled in 6 countries and at 34 study centers. In Part 1, subjects started chemotherapy at day 1 and midostaurin at day 8. In Part 2, subjects started chemotherapy at day 1 and were randomized to midostaurin or placebo at day 8.
Groups:
- Midostaurin: Part 1 (Japan Only): Part 1 was conducted to evaluate the safety and tolerability of midostaurin in combination with daunorubicin/cytarabine induction and high-dose cytarabine consolidation in Japanese patients. The safety evaluation period began on Day 1 of the first induction cycle (Cycle 1 Day 1) and continued until Day 21 of the first consolidation cycle.
- Midostaurin: Part 2: Patients took study drug on day 8-21 during induction and consolidation phase, then on days 1-28 for 12 cycles in the continuation (post-consolidation) phase.
- Placebo: Part 2: Patients took Placebo on day 8 - 21 during induction and consolidation phase, then on days 1-28 for 12 cycles in the continuation (post-consolidation) phase.
Period: Part 1 - Safety Evaluation
Arm/Group | Midostaurin: Part 1 (Japan Only) | Midostaurin: Part 2 | Placebo: Part 2
Started | 5 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 5 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0
Not completed — Disease progression | 1 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0
Period: Part 2 - Efficacy
Arm/Group | Midostaurin: Part 1 (Japan Only) | Midostaurin: Part 2 | Placebo: Part 2
Started (Started = Started Induction phase) | 0 | 30 | 32
Randomized, Not Treated | 0 | 0 | 1
Completed (Completed = Completed Continuation phase) | 0 | 4 | 4
Not Completed | 0 | 26 | 28
Not completed — Adverse Event | 0 | 4 | 6
Not completed — Death | 0 | 3 | 0
Not completed — Physician Decision | 0 | 10 | 16
Not completed — Withdrawal by Subject | 0 | 2 | 1
Not completed — Progressive disease | 0 | 7 | 5

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): The FAS comprised of all subjects to whom study drug (midostaurin/placebo) had been assigned by randomization. Therefore, all Japanese subjects treated during Part 1 were not eligible for the FAS.
Groups:
- Total: Total of all reporting groups
Arm/Group | Midostaurin: Part 1 (Japan Only) | Midostaurin: Part 2 | Placebo: Part 2 | Total
Number analyzed (Participants) | 5 | 30 | 32 | 67
Age, Customized [Number; unit: Participants]
  <60 years | 3 | 27 | 23 | 53
  60 - <65 years | 2 | 2 | 5 | 9
  ≥65 years | 0 | 1 | 4 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 16 | 17 | 35
  Male | 3 | 14 | 15 | 32
Race/Ethnicity, Customized [Number; unit: Participants]
  Japanese | 5 | 12 | 12 | 29
  Korean | 0 | 4 | 6 | 10
  Chinese | 0 | 3 | 10 | 13
  Vietnamese | 0 | 1 | 4 | 5
  Missing | 0 | 1 | 0 | 1
  White | 0 | 9 | 0 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Safety Events (Part 1, Japan Only)
Description: Percentage of Safety Events, defined as death or serious adverse event leading to treatment discontinuation that occurs on or before Day 21 of the first Consolidation cycle. This was determined by the Independent Safety Committee (ISC) to be definitely or probably related to midostaurin. Percentage was calculated based on the percentage of subjects with safety event out of 3 evaluable subjects in Part 1.
Time Frame: up to Day 21 of the first Consolidation cycle; cycle = 28 days
Population: Patients enrolled in Part 1: 3 patients out of 5 patients in Part 1 were evaluable for safety evaluation as determined by Independent Safety Committee (ISC).
Measure: Number; unit: Participants
Arm/Group | Midostaurin: Part 1 (Japan Only) | Midostaurin: Part 2 | Placebo: Part 2
Number analyzed (Participants) | 5 | 0 | 0
Participants
  Experienced at least 1 adverse event (AE) | 5 |  |
  Safety events determined by ISC related to midostaurin (n = 3, 0, 0): number analyzed (Participants) | 3 | 0 | 0
  Safety events determined by ISC related to midostaurin (n = 3, 0, 0) | 0 |  |

2. Primary Outcome: Event Free Survival (EFS) (Part 2 - Randomized, Controlled)
Description: Event Free survival is defined as the time from the date of randomization until an EFS event is observed. An EFS event is defined as a failure to obtain a complete remission (CR) within an induction 2, relapse after CR, or death due to any cause, whichever occurs first.
  The objective was to evaluate the efficacy based on EFS of midostaurin versus placebo in combination with daunorubicin/cytarabine induction, with high-dose cytarabine consolidation, and with midostaurin single agent continuation therapy in newly diagnosed patients with FLT3-mutated AML.
Time Frame: up to 3 years after last patient started treatment
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Midostaurin: Part 2 | Placebo: Part 2
Number analyzed (Participants) | 30 | 32
Months | 7.6 [3.6 to NA] — NA: The final data was not mature to estimate the upper limit of the confidence interval for median EFS. | NA [8.2 to NA] — NA: The Final data was not mature to estimate the median EFS (i.e., not reached) and its upper limit of the confidence interval.
Statistical Analysis 1: Comparison: Midostaurin: Part 2 vs Placebo: Part 2; Test type: Other — Success criteria is considered based on point estimated Hazard ratio; Hazard Ratio, log = 1.326, 95% CI 2-sided [0.624 to 2.818]

3. Secondary Outcome: Overall Survival
Description: Overall survival defined as the time from the date of randomization to date of death due to any cause
Time Frame: up to 3 years after last patient started treatment
Population: FAS: The FAS comprised of all subjects to whom study drug (midostaurin/placebo) had been assigned by randomization. Therefore, all Japanese subjects treated during Part 1 were not eligible for the FAS.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Midostaurin: Part 2 | Placebo: Part 2
Number analyzed (Participants) | 30 | 32
Months | NA [16.8 to NA] — NA: The final data was not mature to estimate the median OS (i.e., not reached) and its upper limit of the confidence interval. | NA [18.8 to NA] — NA: The final data was not mature to estimate the median OS (i.e., not reached) and its upper limit of the confidence interval.

4. Secondary Outcome: Percentage of Participants With Complete Remission (CR)
Description: Complete Remission is defined as the percentage of participants with a CR according to Chelson Criteria, at various timepoints
Time Frame: up to 3 years after last patient started treatment
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Midostaurin: Part 2 | Placebo: Part 2
Number analyzed (Participants) | 30 | 32
Percentage of participants
  Overall CR | 70.0 [50.60 to 85.27] | 78.1 [60.03 to 90.72]
  Morphologic CR with incomplete platelet count recovery (CRp) | 6.7 [0.86 to 22.07] | 0.0 [0.00 to 10.89]
  End of Induction cycle 1 (C1) CR | 56.7 [37.43 to 74.54] | 65.6 [46.81 to 81.43]
  End of Induction C1: Morphologic CRp | 3.3 [0.08 to 17.22] | 0.0 [0.00 to 10.89]
  End of Induction cycle 2 (C2) CR | 13.3 [3.76 to 30.72] | 9.4 [1.98 to 25.02]
  End of Induction C2: Morphologic CRp | 3.3 [0.08 to 17.00] | 0.0 [0.00 to 10.89]
  End of Consolidation CR | 36.7 [19.93 to 56.14] | 43.8 [26.36 to 62.34]
  End of Consolidation Morphologic CRp | 3.3 [0.08 to 17.22] | 9.4 [1.98 to 25.02]
  After treatment discontinuation CR | 10.0 [2.11 to 26.53] | 3.1 [0.08 to 16.22]
  After treatment discontinuation Morphologic CRp | 0.0 [0.00 to 11.57] | 6.3 [0.77 to 20.81]

5. Secondary Outcome: Percentage of Participants With Cumulative Incidence of Relapse (CIR)
Description: CIR (only for patients who achieved CR after study treatment initiation), is measured from the date of first CR to relapse or death due to AML, whichever occurs first.
Time Frame: up to 3 years after last patient started treatment
Population: FAS: The FAS comprised of all subjects to whom study drug (midostaurin/placebo) had been assigned by randomization. Therefore, all Japanese subjects treated during Part 1 were not eligible for the FAS. This analysis was on FAS but only on participants who had achieved a CR.
Measure: Count of Participants; unit: Participants
Arm/Group | Midostaurin: Part 2 | Placebo: Part 2
Number analyzed (Participants) | 30 | 32
Participants | 21 | 25

6. Secondary Outcome: Pharmakinetics (PK) for Midostaurin: AUClast & AUC0-t
Description: Evaluate AUClast & AUC0-t PK parameters for midostaurin. AUClast: The AUC from time zero to the last measurable concentration sampling time (Tlast) (mass x time x volume-1) AUC0-t: The area under the curve (AUC) from time zero to a measurable concentration sampling time (t) (mass x time x volume-1).
Time Frame: Induction Phase: Pre-dose and 1, 3, 6 and 12 hours post dose in Cycle 1 Day 8
Population: PK analysis set for full PK (PAS-full): The PAS-full included all subjects in the PAS-all, who provide an evaluable PK profile. A profile was considered evaluable if all of the following conditions are satisfied: Subject received the planned dose of midostaurin on C1D8 of induction therapy; Subject did not vomit within 4 hours of the dosing of midostaurin on C1D8 of induction therapy; Subject provided at least one primary PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Midostaurin: Part 2
Number analyzed (Participants) | 34
ng*hr/mL
  AUClast | 17900 (53.5)
  AUC0-t: number analyzed (Participants) | 31
  AUC0-t | 19200 (49.0)

7. Secondary Outcome: Pharmakinetics (PK) for Midostaurin: Cmax
Description: Evaluate Cmax parameter for midostaurin. Cmax: The maximum (peak) observed plasma drug concentration after the first dose administration of midostaurin (mass x volume-1).
Time Frame: Induction Phase: Pre-dose and 1, 3, 6 and 12 hours post dose in Cycle 1 Day 8
Population: PAS-full: PK analysis set for full PK (PAS-full): The PAS-full included all subjects in the PAS-all, who provide an evaluable PK profile. A profile was considered evaluable if all of the following conditions are satisfied: Subject received the planned dose of midostaurin on C1D8 of induction therapy; Subject did not vomit within 4 hours of the dosing of midostaurin on C1D8 of induction therapy; Subject provided at least one primary PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Midostaurin: Part 2
Number analyzed (Participants) | 34
ng/mL | 2420 (46.5)

8. Secondary Outcome: Metabolite CGP52421: PK Parameters AUClast, AUC0-t
Description: Evaluate the pharmacokinetic of major metabolite of midostaurin CGP52421. AUClast: The AUC from time zero to the last measurable concentration sampling time (Tlast) (mass x time x volume-1) AUC0-t: The area under the curve (AUC) from time zero to a measurable concentration sampling time (t) (mass x time x volume-1).
Time Frame: Induction Phase: Cycle 1 Day 8
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Midostaurin: Part 2
Number analyzed (Participants) | 34
ng*hr/mL
  AUClast | 754 (116)
  AUC0-t: number analyzed (Participants) | 31
  AUC0-t | 876 (92.3)

9. Secondary Outcome: Metabolite CGP52421: PK Parameter Cmax
Description: Evaluate the pharmacokinetic of major metabolite of midostaurin CGP52421: Cmax. Cmax: The maximum (peak) observed plasma drug concentration after the first dose administration of midostaurin (mass x volume-1).
Time Frame: Induction Phase: Cycle 1 Day 8
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Midostaurin: Part 2
Number analyzed (Participants) | 34
ng/mL | 98.6 (83.5)

10. Secondary Outcome: Metabolite CGP62221: PK Parameters: AUClast, AUC0-t
Description: Evaluate the pharmacokinetic of major metabolite of Midostaurin CGP62221 PK parameters AUClast, AUC0-t
Time Frame: Induction Phase: Cycle 1 Day 8
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Midostaurin: Part 2
Number analyzed (Participants) | 34
ng*hr/mL
  AUClast | 1430 (223)
  AUC0-t: number analyzed (Participants) | 31
  AUC0-t | 1730 (182)

11. Secondary Outcome: Metabolite CGP62221: PK Parameter: Cmax
Description: Evaluate the pharmacokinetic of major metabolite of Midostaurin CGP62221 PK parameter Cmax.
  Cmax: The maximum (peak) observed plasma drug concentration after the first dose administration of midostaurin (mass x volume-1).
Time Frame: Induction Phase: Cycle 1 Day 8
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Midostaurin: Part 2
Number analyzed (Participants) | 34
ng/mL | 196 (159)

12. Secondary Outcome: Change From Baseline in Quality of Life (QoL) Per European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30
Description: The EORTC QLQ-C30 is a 30-item questionnaire with multi-item scales and single-item measures, including five functional scales (physical, role, emotional, cognitive, and social), three symptom scales (fatigue, nausea/vomiting, and pain), six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial impact), and a global health status/QoL scale. Scores range from 0 to 100, with higher scores indicating higher response levels. High functional scale scores denote healthy functioning, high global QoL scores indicate high QoL, and high symptom scores reflect high symptom levels. Scoring follows the EORTC Scoring Manual, reported by absolute change from baseline. EOI = End of Induction; EOCons = End of Consolidation; EOCont = End of Continuation; EOT = End of Treatment.
Time Frame: EOI: up to 1.84 months (after 2 cycles); EOCons: up to 5.52 months (after 4 cycles); EOCont: up to 16.56 months (after 12 cycles); EOT: up to 16.56 months maximum, depending on treatment duration; each cycle = 28 days
Population: Participants in the full analysis set (FAS) with an available assessment for the outcome measure at each timepoint. FAS: The FAS comprised of all subjects to whom study drug (midostaurin/placebo) had been assigned by randomization.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Midostaurin: Part 2 | Placebo: Part 2
Number analyzed (Participants) | 17 | 20
scores on a scale
  EOI: Global health status (GHS):GHS: number analyzed (Participants) | 6 | 3
  EOI: Global health status (GHS):GHS | 27.8 (31.03) | 0.0 (16.67)
  EOCons: GHS:GHS: number analyzed (Participants) | 6 | 11
  EOCons: GHS:GHS | 20.8 (11.49) | 37.1 (24.54)
  EOCont: GHS:GHS: number analyzed (Participants) | 5 | 6
  EOCont: GHS:GHS | 28.3 (22.52) | 27.8 (10.09)
  EOT:GHS:GHS | 25.5 (21.94) | 28.8 (23.33)

13. Secondary Outcome: Quality of Life (QoL) Per Patient Global Impression of Change (PGIC)
Description: The PGIC is a single self-reported item that asks about change in status of subject's overall satisfaction with medication since starting the standalone study. The specific wording of the PGIC is "Directions: Circle the one number that best describes how your overall satisfaction with your medication had changed since starting the study": "Very much improved" =1; "Much improved" =2; "Minimally improved" =3; "No change" =4; "Minimally worse" =5; "Much worse" =6; "Very much worse" =7. PGI-C questions have been widely used to assess the patient perspective of improvement in clinical trials and have shown clinical validity in a variety of indications, including depression, urinary incontinence and adult asthma and the PGIC score determined frequencies and percentages by scheduled timepoint. EOI = End of Induction; EOCons = End of Consolidation; EOCont = End of Continuation; EOT = End of Treatment.
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Number; unit: Participants
Arm/Group | Midostaurin: Part 2 | Placebo: Part 2
Number analyzed (Participants) | 18 | 20
Participants
  EOI: Very much improved | 1 | 0
  EOI: Much improved | 2 | 1
  EOI: Minimally improved | 3 | 0
  EOI: No change | 1 | 1
  EOI: Minimally worse | 0 | 1
  EOCons: Very much improved | 1 | 1
  EOCons: Much improved | 2 | 3
  EOCons: Minimally improved | 2 | 4
  EOCons: No change | 1 | 2
  EOCons: Minimally worse | 0 | 1
  EOCont: Very much improved | 3 | 2
  EOCont: Much improved | 0 | 4
  EOCont: Minimally improved | 1 | 0
  EOCont: No change | 1 | 0
  EOT: Very much improved | 5 | 3
  EOT: Much improved | 4 | 8
  EOT: Minimally improved | 6 | 4
  EOT: No change | 3 | 3
  EOT: Minimally worse | 0 | 2

14. Post Hoc Outcome: All Collected Deaths
Description: Pre-treatment deaths were collected from screening visit up to the first day of treatment, for a maximum duration of 21 days. Participants who died during the screening period are considered as screen failures.
  On-treatment deaths were collected from start of treatment (FPFT) up to 30 days after study drug discontinuation, for a maximum duration of approx. 55 months.
  Post-treatment survival follow-up deaths were collected after the on-treatment period up to approx. 36 months. Participants who did not die during the on-treatment period and had not stopped study participation at the time of data cut-off (when study was terminated) were censored.
Time Frame: Start of study treatment up to 30 days post-treatment for approx. 1 year, prior to study treatment (before randomization) up to LPLV, approx. 55 months
Population: Clinical Database Population: all enrolled participants
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Part 2: Patients took Placebo on day 8 - 21 during induction and consolidation phase, then on days 1-28 for 12 cycles in the continuation (post-consolidation) phase. This group excludes 1 participant who was randomized to placebo but did not receive placebo and died during the on-treatment period.
- Other Participants: These participants were not randomized to any treatment but received chemotherapy and died during the study. This group also includes 1 participant who was randomized to placebo but did not receive placebo and died during the on-treatment period.
Arm/Group | Midostaurin: Part 1 (Japan Only) | Midostaurin: Part 2 | Placebo: Part 2 | Other Participants
Number analyzed (Participants) | 5 | 30 | 31 | 7
Participants
  Total Deaths in study | 3 | 10 | 7 | 7
  Deaths on-treatment | 1 | 3 | 1 | 0
  Post-treatment survival follow-up deaths: number analyzed (Participants) | 4 | 27 | 30 | 7
  Post-treatment survival follow-up deaths | 2 | 7 | 6 | 0
  Deaths - Not randomized to any treatment but received chemotherapy | 0 | 0 | 0 | 6
  Deaths - Randomized to placebo but did not receive drug | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment to 30 days after last dose of study medication (on-treatment), up to approx. 55 months. Deaths were collected in the post-treatment survival follow up from 31 days after last dose of study medication until the end of the study, up to approx. 36 months. These are not considered AEs
Description: An Adverse Event is any sign or symptom occurring during a trial and safety follow-up, excluding deaths in post-treatment survival follow-up. The total at risk includes patients entering post-treatment survival after the 30-day post-treatment period. Death data was reported for all enrolled patients, while Adverse Events data was reported from those receiving at least one dose of the study drug (midostaurin/placebo).
Groups:
- Midostaurin: Part 1 (Japan Only) (On-treatment): Part 1 was conducted to evaluate the safety and tolerability of midostaurin in combination with daunorubicin/cytarabine induction and high-dose cytarabine consolidation in Japanese patients. The safety evaluation period began on Day 1 of the first induction cycle (Cycle 1 Day 1) and continued until Day 21 of the first consolidation cycle.
- Midostaurin: Part 2 (On-treatment): Patients took study drug on day 8-21 during induction and consolidation phase, then on days 1-28 for 12 cycles in the continuation (post-consolidation) phase.
- Placebo Part 2 (On-treatment): Patients took Placebo on day 8 - 21 during induction and consolidation phase, then on days 1-28 for 12 cycles in the continuation (post-consolidation) phase. This group excludes the 1 participant who was randomized to placebo but did not receive placebo and died during the on-treatment period.
- Midostaurin: Part 1 (Japan Only) (Post-treatment Survival Follow-up): Deaths collected in the post- treatment survival follow-up in Part 1 phase (starting from day 31 post- treatment in Part 1). No AEs were collected during this period.
- Midostaurin: Part 2 (Post-treatment Survival Follow-up); Placebo: Part 2 (Post-treatment Survival Follow-up): Deaths collected in the post- treatment survival follow-up phase (starting from day 31 post- treatment). No AEs were collected during this period.
Arm/Group | Midostaurin: Part 1 (Japan Only) (On-treatment) | Midostaurin: Part 2 (On-treatment) | Placebo Part 2 (On-treatment) | Midostaurin: Part 1 (Japan Only) (Post-treatment Survival Follow-up) | Midostaurin: Part 2 (Post-treatment Survival Follow-up) | Placebo: Part 2 (Post-treatment Survival Follow-up) | Other Participants
All-Cause Mortality (participants affected / at risk) | 1/5 | 3/30 | 1/31 | 2/4 | 7/27 | 6/30 | 7/7
Serious Adverse Events (participants affected / at risk) | 2/5 | 12/30 | 10/31 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 5/5 | 30/30 | 31/31 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Midostaurin: Part 1 (Japan Only) (On-treatment) (N=5) | Midostaurin: Part 2 (On-treatment) (N=30) | Placebo Part 2 (On-treatment) (N=31) | Midostaurin: Part 1 (Japan Only) (Post-treatment Survival Follow-up) (N=0) | Midostaurin: Part 2 (Post-treatment Survival Follow-up) (N=0) | Placebo: Part 2 (Post-treatment Survival Follow-up) (N=0) | Other Participants (N=0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 2 | 1 | NA | NA | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | NA | NA | NA | NA
Cardiac failure (Cardiac disorders) | 0 | 1 | 0 | NA | NA | NA | NA
Cardiac failure acute (Cardiac disorders) | 1 | 0 | 0 | NA | NA | NA | NA
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0 | NA | NA | NA | NA
Necrotising colitis (Gastrointestinal disorders) | 0 | 1 | 0 | NA | NA | NA | NA
Proctitis (Gastrointestinal disorders) | 0 | 1 | 0 | NA | NA | NA | NA
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 0 | NA | NA | NA | NA
Pyrexia (General disorders) | 0 | 1 | 2 | NA | NA | NA | NA
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 1 | NA | NA | NA | NA
Candida infection (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA | NA
Escherichia sepsis (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA | NA
Fungaemia (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA | NA
Osteomyelitis (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA | NA
Periodontitis (Infections and infestations) | 0 | 1 | 0 | NA | NA | NA | NA
Pneumonia (Infections and infestations) | 1 | 5 | 2 | NA | NA | NA | NA
Sepsis (Infections and infestations) | 1 | 3 | 1 | NA | NA | NA | NA
Septic shock (Infections and infestations) | 0 | 2 | 1 | NA | NA | NA | NA
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | NA | NA | NA | NA
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | NA | NA | NA | NA
Platelet count decreased (Investigations) | 0 | 0 | 1 | NA | NA | NA | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | NA | NA | NA | NA
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | NA | NA | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 4.99% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Midostaurin: Part 1 (Japan Only) (On-treatment) (N=5) | Midostaurin: Part 2 (On-treatment) (N=30) | Placebo Part 2 (On-treatment) (N=31) | Midostaurin: Part 1 (Japan Only) (Post-treatment Survival Follow-up) (N=0) | Midostaurin: Part 2 (Post-treatment Survival Follow-up) (N=0) | Placebo: Part 2 (Post-treatment Survival Follow-up) (N=0) | Other Participants (N=0)
Anaemia (Blood and lymphatic system disorders) | 3 | 17 | 15 | NA | NA | NA | NA
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 | 2 | NA | NA | NA | NA
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 25 | 21 | NA | NA | NA | NA
Leukopenia (Blood and lymphatic system disorders) | 1 | 2 | 0 | NA | NA | NA | NA
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 2 | 0 | NA | NA | NA | NA
Neutropenia (Blood and lymphatic system disorders) | 1 | 6 | 7 | NA | NA | NA | NA
Pancytopenia (Blood and lymphatic system disorders) | 2 | 1 | 0 | NA | NA | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 10 | 3 | NA | NA | NA | NA
Cardiac failure (Cardiac disorders) | 1 | 1 | 0 | NA | NA | NA | NA
Cardiac hypertrophy (Cardiac disorders) | 1 | 0 | 0 | NA | NA | NA | NA
Supraventricular tachycardia (Cardiac disorders) | 2 | 0 | 0 | NA | NA | NA | NA
Tachycardia (Cardiac disorders) | 1 | 1 | 0 | NA | NA | NA | NA
Dry eye (Eye disorders) | 0 | 2 | 2 | NA | NA | NA | NA
Eye pain (Eye disorders) | 0 | 1 | 2 | NA | NA | NA | NA
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 2 | NA | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | 2 | 3 | 6 | NA | NA | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 1 | 10 | 4 | NA | NA | NA | NA
Constipation (Gastrointestinal disorders) | 1 | 10 | 14 | NA | NA | NA | NA
Dental caries (Gastrointestinal disorders) | 1 | 1 | 2 | NA | NA | NA | NA
Diarrhoea (Gastrointestinal disorders) | 2 | 20 | 17 | NA | NA | NA | NA
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 2 | NA | NA | NA | NA
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 2 | 0 | NA | NA | NA | NA
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2 | NA | NA | NA | NA
Gastrointestinal mucosal disorder (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA | NA
Gingival bleeding (Gastrointestinal disorders) | 0 | 2 | 2 | NA | NA | NA | NA
Gingival pain (Gastrointestinal disorders) | 0 | 3 | 2 | NA | NA | NA | NA
Haemorrhoids (Gastrointestinal disorders) | 1 | 5 | 3 | NA | NA | NA | NA
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA | NA
Mouth ulceration (Gastrointestinal disorders) | 1 | 1 | 3 | NA | NA | NA | NA
Nausea (Gastrointestinal disorders) | 5 | 17 | 17 | NA | NA | NA | NA
Neutropenic colitis (Gastrointestinal disorders) | 0 | 2 | 0 | NA | NA | NA | NA
Proctalgia (Gastrointestinal disorders) | 0 | 3 | 2 | NA | NA | NA | NA
Stomatitis (Gastrointestinal disorders) | 3 | 9 | 10 | NA | NA | NA | NA
Toothache (Gastrointestinal disorders) | 1 | 0 | 1 | NA | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 3 | 8 | 14 | NA | NA | NA | NA
Asthenia (General disorders) | 0 | 3 | 0 | NA | NA | NA | NA
Catheter site erythema (General disorders) | 1 | 0 | 0 | NA | NA | NA | NA
Catheter site pain (General disorders) | 1 | 0 | 0 | NA | NA | NA | NA
Fatigue (General disorders) | 0 | 1 | 2 | NA | NA | NA | NA
Generalised oedema (General disorders) | 0 | 2 | 4 | NA | NA | NA | NA
Malaise (General disorders) | 4 | 3 | 2 | NA | NA | NA | NA
Oedema (General disorders) | 0 | 2 | 1 | NA | NA | NA | NA
Oedema peripheral (General disorders) | 0 | 2 | 3 | NA | NA | NA | NA
Pain (General disorders) | 1 | 0 | 2 | NA | NA | NA | NA
Pyrexia (General disorders) | 4 | 13 | 19 | NA | NA | NA | NA
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0 | NA | NA | NA | NA
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 2 | 3 | NA | NA | NA | NA
Hypersensitivity (Immune system disorders) | 2 | 1 | 0 | NA | NA | NA | NA
Bacteraemia (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA | NA
Bronchitis (Infections and infestations) | 1 | 1 | 0 | NA | NA | NA | NA
Catheter site cellulitis (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA | NA
Cellulitis (Infections and infestations) | 0 | 2 | 1 | NA | NA | NA | NA
Cellulitis of male external genital organ (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA | NA
Clostridium difficile colitis (Infections and infestations) | 2 | 1 | 0 | NA | NA | NA | NA
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 3 | NA | NA | NA | NA
Conjunctivitis (Infections and infestations) | 0 | 0 | 2 | NA | NA | NA | NA
Device related infection (Infections and infestations) | 1 | 2 | 3 | NA | NA | NA | NA
Ecthyma (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA | NA
Enterocolitis infectious (Infections and infestations) | 0 | 2 | 0 | NA | NA | NA | NA
Escherichia bacteraemia (Infections and infestations) | 0 | 1 | 2 | NA | NA | NA | NA
Gingivitis (Infections and infestations) | 1 | 3 | 1 | NA | NA | NA | NA
Hepatosplenic candidiasis (Infections and infestations) | 0 | 2 | 0 | NA | NA | NA | NA
Herpes zoster (Infections and infestations) | 0 | 1 | 2 | NA | NA | NA | NA
Periodontitis (Infections and infestations) | 0 | 2 | 3 | NA | NA | NA | NA
Pharyngitis (Infections and infestations) | 1 | 2 | 0 | NA | NA | NA | NA
Pneumonia (Infections and infestations) | 1 | 6 | 7 | NA | NA | NA | NA
Pneumonia fungal (Infections and infestations) | 0 | 2 | 1 | NA | NA | NA | NA
Sepsis (Infections and infestations) | 0 | 4 | 3 | NA | NA | NA | NA
Sinusitis (Infections and infestations) | 1 | 0 | 1 | NA | NA | NA | NA
Skin infection (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA | NA
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 3 | NA | NA | NA | NA
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1 | 2 | NA | NA | NA | NA
Fall (Injury, poisoning and procedural complications) | 1 | 2 | 0 | NA | NA | NA | NA
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 2 | NA | NA | NA | NA
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1 | 1 | NA | NA | NA | NA
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 2 | 5 | NA | NA | NA | NA
Wound complication (Injury, poisoning and procedural complications) | 0 | 2 | 0 | NA | NA | NA | NA
Alanine aminotransferase increased (Investigations) | 1 | 11 | 7 | NA | NA | NA | NA
Amylase increased (Investigations) | 1 | 1 | 2 | NA | NA | NA | NA
Antithrombin III decreased (Investigations) | 1 | 0 | 0 | NA | NA | NA | NA
Aspartate aminotransferase increased (Investigations) | 2 | 6 | 5 | NA | NA | NA | NA
Blood alkaline phosphatase increased (Investigations) | 0 | 2 | 2 | NA | NA | NA | NA
Blood bilirubin increased (Investigations) | 1 | 2 | 5 | NA | NA | NA | NA
Blood creatinine increased (Investigations) | 0 | 2 | 0 | NA | NA | NA | NA
Coagulation test abnormal (Investigations) | 1 | 0 | 0 | NA | NA | NA | NA
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 2 | NA | NA | NA | NA
Full blood count increased (Investigations) | 1 | 0 | 0 | NA | NA | NA | NA
Gamma-glutamyltransferase increased (Investigations) | 1 | 4 | 1 | NA | NA | NA | NA
Immunoglobulins decreased (Investigations) | 1 | 0 | 0 | NA | NA | NA | NA
Lymphocyte count decreased (Investigations) | 0 | 1 | 3 | NA | NA | NA | NA
Neutrophil count decreased (Investigations) | 1 | 11 | 16 | NA | NA | NA | NA
Platelet count decreased (Investigations) | 1 | 14 | 18 | NA | NA | NA | NA
Ventilation/perfusion scan abnormal (Investigations) | 1 | 0 | 0 | NA | NA | NA | NA
Weight decreased (Investigations) | 0 | 6 | 7 | NA | NA | NA | NA
Weight increased (Investigations) | 0 | 0 | 2 | NA | NA | NA | NA
White blood cell count decreased (Investigations) | 0 | 11 | 15 | NA | NA | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 3 | 6 | 7 | NA | NA | NA | NA
Fluid retention (Metabolism and nutrition disorders) | 0 | 3 | 0 | NA | NA | NA | NA
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | NA | NA | NA | NA
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 2 | 1 | NA | NA | NA | NA
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | NA | NA | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 7 | 11 | NA | NA | NA | NA
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2 | 3 | NA | NA | NA | NA
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | NA | NA | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 3 | NA | NA | NA | NA
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | NA | NA | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 4 | 4 | NA | NA | NA | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 4 | NA | NA | NA | NA
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | NA | NA | NA | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | NA | NA | NA | NA
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | NA | NA | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3 | NA | NA | NA | NA
Dizziness (Nervous system disorders) | 0 | 3 | 0 | NA | NA | NA | NA
Dysgeusia (Nervous system disorders) | 1 | 3 | 1 | NA | NA | NA | NA
Head discomfort (Nervous system disorders) | 1 | 0 | 0 | NA | NA | NA | NA
Headache (Nervous system disorders) | 3 | 8 | 8 | NA | NA | NA | NA
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 2 | NA | NA | NA | NA
Presyncope (Nervous system disorders) | 1 | 0 | 2 | NA | NA | NA | NA
Delirium (Psychiatric disorders) | 1 | 0 | 0 | NA | NA | NA | NA
Insomnia (Psychiatric disorders) | 1 | 5 | 10 | NA | NA | NA | NA
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0 | NA | NA | NA | NA
Haematuria (Renal and urinary disorders) | 0 | 2 | 3 | NA | NA | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 8 | NA | NA | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | NA | NA | NA | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | NA | NA | NA | NA
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | NA | NA | NA | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA | NA | NA | NA
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 5 | NA | NA | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | NA | NA | NA | NA
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | NA | NA | NA | NA
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA | NA | NA | NA
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | NA | NA | NA | NA
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 7 | 3 | NA | NA | NA | NA
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 3 | 3 | NA | NA | NA | NA
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | NA | NA | NA | NA
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | NA | NA | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 5 | 4 | NA | NA | NA | NA
Rash (Skin and subcutaneous tissue disorders) | 2 | 10 | 18 | NA | NA | NA | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | NA | NA | NA | NA
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | NA | NA | NA | NA
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 8 | 3 | NA | NA | NA | NA
Flushing (Vascular disorders) | 1 | 0 | 0 | NA | NA | NA | NA
Haematoma (Vascular disorders) | 0 | 2 | 0 | NA | NA | NA | NA
Hypertension (Vascular disorders) | 0 | 3 | 0 | NA | NA | NA | NA
Hypotension (Vascular disorders) | 0 | 2 | 4 | NA | NA | NA | NA
Phlebitis (Vascular disorders) | 0 | 0 | 2 | NA | NA | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2020-09-10): https://cdn.clinicaltrials.gov/large-docs/30/NCT03280030/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-06): https://cdn.clinicaltrials.gov/large-docs/30/NCT03280030/SAP_001.pdf